CLINICAL TRIAL: NCT05982028
Title: Evaluation of Patients' Quality of Life and Treatment Outcomes After Pilonidal Cyst Operations.
Brief Title: Patients' Quality of Life After Pilonidal Cyst Operations.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Edvinas Dainius, Principal Investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PC1 - 4
Record Dates: First submitted 2023-07-15; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Pilonidal Cyst; Pain Postoperative; Quality of Life
MeSH Terms: conditions — Pilonidal Sinus; Pain, Postoperative | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pit picking group (Experimental): Minimally invasive pilonidal cyst surgery.
  Interventions: Procedure: Minimally invasive pit-picking surgery
- Excision group (Experimental): Radical surgical pilonidal cyst excision without suturing
  Interventions: Procedure: Radical surgical excision without suturing

INTERVENTIONS:
Procedure: Minimally invasive pit-picking surgery — Midline pits and secondary fistula openings were probed to determine the direction and length of any associated sinus tracts, followed by an excision with a 3 or 5 mm punch biopsy needle, depending on the size of the pit. A 2 cm lateral incision was made parallel to the pilonidal cyst. Hair and granulations within the sinus tracts were removed, and the cyst cavity was drained through the incision. Nonabsorbable monofilament sutures were used to close the excisional wounds of the pits and secondary fistula. Once haemostasis was achieved, the wound was covered with a sterile gauze with 10 % povidone-iodine solution.
  Arms: Pit picking group
Procedure: Radical surgical excision without suturing — Under the guidance of brilliant green, the cavity of the pilonidal cyst, along with the sinus tracts and fistulas, was marked. A symmetric elliptical incision was made to excise the pits and secondary fistula openings. The pilonidal cyst was removed from the healthy subcutaneous tissue and sacrococcygeal fascia using monopolar electrocautery. The wound was not sutured and was left open to heal by secondary intention. After haemostasis was achieved, the wound was covered with sterile gauze with 10 % povidone-iodine solution.
  Arms: Excision group

SUMMARY:
Biomedical research consists of two main parts. In the first part, the pilonidal cyst-specific quality of life questionnaire is compiled, adapted, validated, tested for suitability in assessing patients after pilonidal cyst operations.

The second part will compare two pilonidal cyst operations. A prospective, comparative, randomized clinical study will be conducted.

DETAILED DESCRIPTION:
The first part includes the creation, adaptation, validity and suitability of the pilonidal cyst-specific quality of life questionnaire in assessing patients after pilonidal cyst operations, verification and evaluation of the quality of life and its dynamics after these operations. A survey of patients operated on for acute and chronic pilonidal cysts will be conducted. The main evaluation criteria of the first part will be the internal consistency of the questionnaire, the stability of the measurements, the construct validity and the frequency of patients with moderate and severe symptoms according to the specific quality of life questionnaire after pilonidal cyst surgery and the SF36v2 quality of life questionnaire.

The second part will compare two pilonidal cyst operations. A prospective, comparative, randomized clinical study will be conducted. This part of the study will study patients scheduled for surgery for chronic pilonidal cyst. Patients will be randomized into two groups, a group that will undergo radical excision of the pilonidal cyst without suturing the wound and a group that will undergo minimally invasive "pit picking" surgery. Patients will be interviewed before surgery, as well as on the first and second day after surgery. Discharged patients will complete quality-of-life questionnaires at 1, 2 weeks, and 2 months. Patients will be invited for a visit after 1 and 6 months, wound healing, disease recurrence and quality of life will be evaluated. The main evaluation criteria of the second part will be objective data - postoperative complications, wound healing time, duration of incapacity for work, frequency of disease recurrence and subjective data - changes in pain (VAS 10 cm scale) and quality of life total points according to SF36v2 and the specific life questionnaire created after radical pilonidal cyst excision and "pit picking" operations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 (men and women)
2. Chronic symptomatic (primary or recurrent) pilonidal cyst
3. American Society of Anesthesiologists physical status I to III
4. Signed the person's information and consent form to participate in the study.

Exclusion Criteria:

1. Acute pilonidal cyst
2. Patients who do not speak Lithuanian
3. Cognitive, visual, auditory and locomotor system disorders
4. Insufficiency of kidneys, liver, cardiopulmonary system
5. Refuses to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain after surgery | One week after surgery
  Postoperative pain will be assessed on a VAS 100 mm scale. Patients will mark their pain at rest on a specified 100 mm scale at the specified time.

SECONDARY OUTCOMES:
Rate of disease recurrence | Recurrence will be assessed 6 months and 2 years after surgery
  Disease recurrence will be assessed by clinical examination.
Pain after surgery | One day after surgery
  Postoperative pain will be assessed on a VAS 100 mm scale. Patients will mark their pain
Pain after surgery | Two days after surgery
  Postoperative pain will be assessed on a VAS 100 mm scale. Patients will mark their pain
Pain after surgery | Two weeks after surgery
  Postoperative pain will be assessed on a VAS 100 mm scale. Patients will mark their pain
Pain after surgery | One month after surgery
  Postoperative pain will be assessed on a VAS 100 mm scale. Patients will mark their pain
Pain after surgery | Two months after surgery
  Postoperative pain will be assessed on a VAS 100 mm scale. Patients will mark their pain
Pain after surgery | Six months after surgery
  Postoperative pain will be assessed on a VAS 100 mm scale. Patients will mark their pain

OTHER OUTCOMES:
Postoperative complications | 1 months after surgery
  Patients will report past complications.
Quality of life according to the 36-Item Short Form Survey (SF-36). | Before surgery, 1 and 2 days after surgery, 1 and 2 weeks after surgery, 1, 2 and 6 months after surgery. Change from baseline in quality of life scores over a 6-month period will be assessed.
  Patients fill out the the 36-Item Short Form Survey (SF-36). All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible. Aggregate scores are compiled as a percentage of the total points possible, using the RAND scoring table. The scores from those questions that address each specific area of functional health status are then averaged together, for a final score within each of the 8 dimensions measured (physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/ fatigue, emotional well being, social functioning, pain, general health). All 8 categories are scored in the same way.
Duration of disability | 1 month after surgery
  Patients will note the duration of incapacity for work.
Wound healing time | Six months after surgery
  Patients will note the time when the wound healed.
Quality of life total scores according to a specific life questionnaire developed by the researcher. | Before surgery, 1 and 2 days after surgery, 1 and 2 weeks after surgery, 1, 2 and 6 months after surgery. Change from baseline in quality of life scores over a 6-month period will be assessed.
  Patients fill out a specific life questionnaire. This questionnaire consists of 20 questions, the value of each question is from 1 to 5 points. The minimum score value is 20, the maximum score value is 100. A lower score value indicates a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Clinic of General Surgery, Kaunas, Lithuania